CLINICAL TRIAL: NCT04810156
Title: A National Prospective Study of Patients With Hepatitis Induced by Immune Checkpoint Inhibitors; Characterization of Liver Injury, Outcome of Therapy and Randomization to Either Prednisolone or Mycophenolate Mofetil Treatment in Case of Relapse
Brief Title: Treatment Efficacy of Corticosteroids and Mycophenolate Mofetil in Patients With Immune Related Hepatitis
Acronym: I-HEP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, M.D. Professor, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA2032
Record Dates: First submitted 2021-03-17; First posted 2021-03-22 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Hepatitis, Drug-Induced
Keywords: Hepatitis; Immunotherapy; Cancer; Adverse events; Immune checkpoint inhibitors; Steroid-refractory; Steroid-dependent
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Hepatitis; Neoplasms | interventions — Mycophenolic Acid; Methylprednisolone Hemisuccinate; Methylprednisolone; Adrenal Cortex Hormones; Steroids; Ursodeoxycholic Acid; Prednisone

STUDY DESIGN:
Intervention Model Description: The aim is to enroll around 40 patients in Cohort A for prospectively characterize the various patterns of liver injury histopathologically, biochemically, and phenotypically that are induced by ICI, and the response to treatment (steroids and MMF).
  Cohort B: 20 patients who experienced a relapse of ir-hepatitis (grade ≥2) during prednisolone tapering or within one month after ended tapering will be randomized to either 100% dose of current steroid dose or restart of steroid 0.5-1 mg/kg versus adding MMF (if the patient received prednisolone the tapering plan hereof is continued, prednisolone up to 25 mg can be added if clinical indicated). Treatment efficacy is evaluated after seven days, if sufficient response the patients continued treatment, in case of insufficient response a cross-over will be performed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A: Steroids and MMF in grade 3-4 ir-hepatitis (Active Comparator): Patients with ≥ 3 grade ir-hepatitis will be treated with high-dose steroids 2 mg/kg/day intravenously. A diagnostic liver biopsy will be taken. Patients with mixed or cholestatic liver injury patterns will be added UDCA. Treatment evaluation will be performed after 72 hours, patients in UDCA will be evaluated will be on day 7. Patients with sufficient steroid response defined as ≥ 20% reduction in ALT, AST, ALP or bilirubin at day 4 or day 7 will undergo steroid tapering with a transition to peroral steroids. Patients with initial insufficient treatment response, defined as less than < 20% reduction in ALT, AST, ALP, or bilirubin, are considered as having a steroid-refractory condition and will be added MMF. In case of no response or increase of ALT, AST, ALP, or bilirubin during treatment with steroids plus MMF a third-line treatment may be introduced according to the individual treating hepatologist.
  Interventions: Drug: Mycophenolate Mofetil; Drug: Solu-Medrol; Drug: Ursodeoxycholic acid; Drug: Prednisone tablet
- Cohort B: Prednisolone versus MMF in steroiddependent ≥2 ir-hepatitis (randomized) (Active Comparator): Patients who experienced relapse of ir-hepatitis of grade ≥2 during prednisolone tapering or within one months after ended tapering will be randomized to either 100% dose of current steroid dose or restart of steroid 0.5-1 mg/kg versus adding MMF (if the patient received prednisolone the tapering plan hereof is continued, prednisolone up to 25 mg can be added if clinical indicated). Treatment efficacy is evaluated after seven days, if sufficient response the patients continued treatment, in case of insufficient response a cross-over will be performed.
  Interventions: Drug: Mycophenolate Mofetil; Drug: Ursodeoxycholic acid; Drug: Prednisone tablet

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Day 1: MMF 500 mg twice a day Day 2: MMF 1000 mg twice a day
  Other Names: Cellcept; Myfenax
Drug: Solu-Medrol — 2 mg/kg/day
  Other Names: Methylprednisolone; Medrol; Corticosteroids; Steroid
  Arms: Cohort A: Steroids and MMF in grade 3-4 ir-hepatitis
Drug: Ursodeoxycholic acid — Patients with mixed or cholestatic liver injury pattern will also be administrated peroral UDCA according to weight
  Other Names: ursochol
Drug: Prednisone tablet — Shift from solu-medrol IV to peroral prednisolon. A tapering plan will be performed.
  Other Names: steroid; Corticosteroids

SUMMARY:
This clinical trial is to clarify and investigate the patterns of immune-related hepatitis and the optimal treatment choice for patients who are steroid-dependent. The project aims to prospectively characterize the various histopathological, biochemical, and phenotypical liver injury patterns induced by immune checkpoint inhibitors and the treatment responses to corticosteroids. Furthermore, the effect of adding a second-line immunosuppressive drug, either MMF in steroid-refractory or steroid-dependent cases will be explored and compared.

DETAILED DESCRIPTION:
The number of patients treated with immune checkpoint inhibitors (ICI) is expanding worldwide due to an increasing number of indications, including additional types of cancer, combination of ICI with other antineoplastic therapies and have recently moved into the adjuvant setting. According to clinical trial material, almost all patients in ICI treatment will eventually develop any grade of an adverse event, here, estimated in up to 90 percent of treated patients. Around 10-30 percent of ICI-treated patients will show signs of liver injury related to ICI treatment and will be diagnosed with immune-related hepatitis. The treatment hereof should include observation and medium-dose steroids in low-grade asymptomatic patients (grade ≤ 2 ir-hepatitis) and high-dose steroids in higher grades according to the current European and American guidelines. However, up to 25 percent of patients with ir-hepatitis may not respond properly to steroids due to primary resistance or relapse during tapering. These patients should be offered a second-line immunosuppressive treatment. The present recommendation for patients with steroid-dependent ir-hepatitis is based on the case series and includes immunosuppressive treatment with mycophenolate mofetil (MMF). To date, no evidence exists for which second-line treatment to choose.

However, in the clinic, the initiation of MMF may be delayed, meanwhile, patients are typically treated with an increased dose of steroids. In some cases, an increased dose of steroids with prolonged tapering can be sufficient. We want to explore if increased doses of steroids or adding MMF is the best strategy for relapse of hepatitis.

In addition, patients with signs of biliary or mixed liver injury may benefit from adding ursodeoxycholic acid (UDCA).

ELIGIBILITY:
Inclusion Criteria:

Cohort A:

- Abnormal liver parameters equal to ≥ grade 3 ir-hepatitis defined as; AST/ALT/ALP >5 x ULN, INR ≥ 2.5 x ULN, or bilirubin > 3.0 x ULN

Cohort B:

- Patients who recur during or within one months of prednisolone tapering of ≥2 ir-hepatitis equal to AST/ALT ≥3 x ULN, ALP ≥2.5 x ULN, INR ≥ 1.5 x ULN, or bilirubin ≥ 3.0 x ULN

Cohort A and Cohort B

* Histologically confirmed solid cancer
* Treatment with cytotoxic T-lymphocyte-associated protein-4 (CTLA-4) or Programmed Cell Death-1 (PD-1)/Programmed Cell Death Ligand-1 (PD-L1) inhibitor or a combination of CTLA-4 plus PD-1 inhibitors within 6 months
* Age: ≥ 18 years
* Women of childbearing potential: Negative serum pregnancy test and must use effective contraception. This applies from screening and until 6 months after treatment. Birth control pills, spiral, depot injection with gestagen, subdermal implantation, hormonal vaginal ring and transdermal depot patch are all considered effective contraceptives
* Men with female partner of childbearing potential must use effective contraception from screening and until 6 months after treatment. Effective contraceptives are as described above for the female partner. In addition, documented vasectomy and sterility or double barrier contraception are considered effective contraceptives
* Signed statement of consent after receiving oral and written study information
* Willingness to participate in the planned treatment and follow-up and capable of handling toxicities.

Exclusion Criteria:

* Concomitant chemotherapy treatment or tyrosine kinases or angiogenesis inhibitors
* Concomitant immunosuppressive medication except prednisolone
* Patients with hepatocellular carcinoma
* Known hypersensitivity to one of the active drugs or excipients
* Uncontrolled infection
* Acute viral hepatitis
* Any medical condition that will interfere with patient compliance or safety
* Simultaneous treatment with other experimental drugs or other anticancer drugs
* Pregnant or breastfeeding females
* Phenylketonuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-07 (Actual); Primary Completion 2025-04-07 (Estimated); Study Completion 2025-11-07 (Estimated)

PRIMARY OUTCOMES:
Treatment-assessed hepatitis response rates | Through study completion, an average of 5 years
  Treatment-assessed hepatitis response rates with steroids and steroids plus either mycophenolate mofetil or tacrolimus
Time to response or downgrading of liver injury in days | Until completion of the study, an average of 5 years
  Time to response or downgrading of liver injury in patients with ≥grade 3 ir-hepatitis measured as; Days to ≥20 percent reduction in liver specific transaminases (ALT/AST) or bilirubin Days to shift to peroral prednisolone and discharge

SECONDARY OUTCOMES:
Relapse rate of immune related hepatitis ≥2 during tapering plan | Through study completion, an average of 5 years
  Percent of patients with relapse to grade ≥2 hepatitis during steroid or during steroid plus either mycophenolate mofetil or tacrolimus tapering.
Time to downgrading of hepatotoxicity assessed by CTCAE v5.0 | Through study completion, an average of 5 years
  Time to downgrading of hepatotoxicity from grade 4 to grade 3, to grade 2 and to grade 1, respectively, assessed by CTCAE v5.0
Description of histopathological changes in liver tissue | Until completion of the study, an average of 5 years
  Number of patients with hepatocellular, cholestatic and mixed liver injury respectively, assessed by histological findings of predominant injury to hepatocytes, bile ducts or combined.
Incidence of abnormal laboratory test results | Until completion of the study, an average of 5 years
  Incidence of abnormal laboratory test results in blood
Cumulated doses of corticosteroids and MMF respectively | Until completion of the study, an average of 5 years
  Cumulated doses of corticosteroids and MMF respectively, during the study period of 6 months
Cancer progression free survival at 6 months | Until completion of the study, an average of 5 years
  Cancer progression free survival at 6 months
Overall survival rates at 6 months | Until completion of the study, an average of 5 years
  Overall survival rates at 6 months

OTHER OUTCOMES:
Blood biomarkers | Until completion of the study, an average of 5 years
  Correlation of the baseline immune markers, genomics and other biomarkers in blood
Description of changes in the fecal microbiome | Until completion of the study, an average of 5 years
  Description of changes in the fecal microbiome and characterization of the prevalence of specific bacteria e.g. Faecalibacterium and Firmicutes

CONTACTS AND LOCATIONS:
Overall Officials: Inge M Svane, Study Director — Study Director, National Center for Cancer Immune Therapy, Dept. of Oncology, Hospital Herlev; Rikke B Holmstrøm, Principal Investigator — Ph.D student, National Center for Cancer Immune Therapy, Dept. of Oncology, Hospital Herlev
Locations (5):
- Denmark (5):
  - Herlev University Hospital, Herlev, Copenhagen
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense